CLINICAL TRIAL: NCT00464685
Title: Safety and Efficacy of a New Treatment in Combination With Laser for Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 206207-012
Record Dates: First submitted 2007-04-20; First posted 2007-04-24 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 700 µg Dexamethasone Implant and Laser Photocoagulation (Experimental): Initial intravitreal injection of 700 µg dexamethasone with up to 1 additional treatment based on re-treatment criteria. Initial laser photocoagulation with up to 3 additional treatments based on re-treatment criteria.
  Interventions: Drug: Dexamethasone; Procedure: Laser Photocoagulation
- Sham Implant and Laser Photocoagulation (Sham Comparator): Initial sham injection with up to 1 additional treatment based on re-treatment criteria. Initial laser photocoagulation with up to 3 additional treatments based on re-treatment criteria.
  Interventions: Drug: Sham injection; Procedure: Laser Photocoagulation

INTERVENTIONS:
Drug: Dexamethasone — Initial intravitreal injection of 700 µg dexamethasone with up to 1 additional treatment based on re-treatment criteria.
  Other Names: Posurdex®
  Arms: 700 µg Dexamethasone Implant and Laser Photocoagulation
Drug: Sham injection — Initial sham injection with up to 1 additional treatment based on re-treatment criteria.
  Arms: Sham Implant and Laser Photocoagulation
Procedure: Laser Photocoagulation — Initial laser photocoagulation with up to 3 additional treatments based on re-treatment criteria.

SUMMARY:
This study will evaluate the safety and efficacy of the intravitreal implant of dexamethasone with laser treatment vs. laser treatment alone in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with diabetic macular edema
* Decrease in visual acuity in at least one eye as a result of macular edema (20/50 or worse)
* Visual acuity in other eye no worse than 20/200

Exclusion Criteria:

* Known anticipated need for ocular surgery within next 12 months
* History of glaucoma or current high eye pressure requiring more than 1 medication
* Uncontrolled systemic disease
* Known steroid-responder
* Use of systemic steroids - Use of Warfarin/Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2010-02-08 (Actual); Study Completion 2010-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Artesia, California, United States
- Victoria, British Columbia, Canada

REFERENCES:
- [Background] Callanan DG, Gupta S, Boyer DS, Ciulla TA, Singer MA, Kuppermann BD, Liu CC, Li XY, Hollander DA, Schiffman RM, Whitcup SM; Ozurdex PLACID Study Group. Dexamethasone intravitreal implant in combination with laser photocoagulation for the treatment of diffuse diabetic macular edema. Ophthalmology. 2013 Sep;120(9):1843-51. doi: 10.1016/j.ophtha.2013.02.018. Epub 2013 May 22. PMID 23706947

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Started | 126 | 127
Completed | 103 | 94
Not Completed | 23 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation | Total
Number analyzed (Participants) | 126 | 127 | 253
Age, Customized [Number; unit: Participants]
  <45 years | 7 | 3 | 10
  45 to 65 years | 72 | 84 | 156
  >65 years | 47 | 40 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 125
  Male | 62 | 66 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least 10 Letters of Improvement in Best Corrected Visual Acuity (BCVA) From Baseline in the Study Eye
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates improvement and a decrease in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Month 12
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Number analyzed (Participants) | 126 | 127
Percentage of Patients | 27.8 | 23.6

2. Secondary Outcome: Change From Baseline in BCVA in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Number analyzed (Participants) | 126 | 127
Letters Read Correctly
  Baseline | 57.6 (9.38) | 57.8 (9.66)
  Change from Baseline at Month 12 | 2.9 (11.45) | 2.1 (12.05)

3. Secondary Outcome: Change From Baseline in Central Subfield Retinal Thickness in the Study Eye
Description: Central subfield retinal thickness is assessed in the study eye by Optical Coherence Tomography (OCT). The central subfield is an area in the retina (back of the eye). OCT is a laser-based, noninvasive, diagnostic system that provides high-resolution, three-dimensional images of the retina from which retinal thickness can be measured. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Month 12
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Number analyzed (Participants) | 126 | 127
Microns
  Baseline | 438.4 (133.93) | 430.3 (131.15)
  Change from Baseline at Month 12 | -102.8 (130.86) | -125.3 (123.38)

4. Secondary Outcome: Change From Baseline in the Focal Leakage Area in the Study Eye
Description: Focal leakage area in the study eye is assessed using fluorescein angiography. A positive number change from baseline indicates a worsening and a negative number change from baseline indicates an improvement.
Time Frame: Baseline, Month 12
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Millimeters Squared (mm^2)
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Number analyzed (Participants) | 126 | 127
Millimeters Squared (mm^2)
  Baseline | 0.6 (1.46) | 1.1 (2.64)
  Change from Baseline at Month 12 | -0.2 (0.96) | -0.7 (3.07)

5. Secondary Outcome: Time to Retreatment in the Study Eye
Description: Time to retreatment in the study eye is defined as the number of days between the initial treatment and re-treatment with the study medication.
Time Frame: 12 Months
Population: Intent to Treat: all randomized patients
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Number analyzed (Participants) | 126 | 127
Days | 189 [189 to 197] | 196 [189 to 216]

ADVERSE EVENTS:
Description: The Safety Population was used to assess all serious adverse events (SAEs) and adverse events (AEs) and included all patients who were randomized and treated.
Arm/Group | 700 µg Dexamethasone Implant and Laser Photocoagulation | Sham Implant and Laser Photocoagulation
Serious Adverse Events (participants affected / at risk) | 23/125 | 27/127
Other Adverse Events (participants affected / at risk) | 125/125 | 127/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone Implant and Laser Photocoagulation (N=125) | Sham Implant and Laser Photocoagulation (N=127)
Pneumonia (Infections and infestations) | 2 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 0
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal Failure (Renal and urinary disorders) | 1 | 1
Aortic Stenosis (Vascular disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Diabetic Foot Infection (Infections and infestations) | 1 | 0
Dialysis Disequilibrium Syndrome (Injury, poisoning and procedural complications) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoglycaemic Seizure (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0
Gangrene (Infections and infestations) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardio-respiratory Arrest (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal Necrosis (Gastrointestinal disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Incision Site Infection (Infections and infestations) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone Implant and Laser Photocoagulation (N=125) | Sham Implant and Laser Photocoagulation (N=127)
Conjunctival Haemorrhage (Eye disorders) | 27 | 24
Vitreous Haemorrhage (Eye disorders) | 17 | 10
Visual Acuity Reduced (Eye disorders) | 14 | 18
Cataract (Eye disorders) | 14 | 8
Eye Pain (Eye disorders) | 13 | 11
Vitreous Floaters (Eye disorders) | 13 | 10
Macular Oedema (Eye disorders) | 11 | 9
Maculopathy (Eye disorders) | 9 | 8
Vitreous Detachment (Eye disorders) | 9 | 3
Retinal Exudates (Eye disorders) | 8 | 7
Diabetic Retinal Oedema (Eye disorders) | 7 | 11
Retinal Haemorrhage (Eye disorders) | 7 | 8
Vision Blurred (Eye disorders) | 7 | 8
Oedema Peripheral (General disorders) | 3 | 8
Bronchitis (Infections and infestations) | 8 | 5
Upper Respiratory Infection (Infections and infestations) | 5 | 7
Intraocular Pressure Increased (Investigations) | 28 | 8
Headache (Nervous system disorders) | 3 | 9
Hypertension (Vascular disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.